CLINICAL TRIAL: NCT00127933
Title: An Open-label Study of Xeloda Plus Taxotere on Treatment Response in Patients With HER2-neu-negative, and the Addition of Herceptin for HER2-neu-positive Breast Cancer
Brief Title: XeNA Study - A Study of Xeloda (Capecitabine) in Patients With Invasive Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18530
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Docetaxel; Trastuzumab

ARMS (2):
- HER2-NEU Positive (Experimental)
  Interventions: Drug: capecitabine [Xeloda]; Drug: Taxotere; Drug: Herceptin (HER2-neu positive patients only)
- HER2-NEU Negative (Experimental)
  Interventions: Drug: capecitabine [Xeloda]; Drug: Taxotere

INTERVENTIONS:
Drug: capecitabine [Xeloda] — 825mg/m2 po bid on days 1-14 of each 3 week cycle
  Arms: HER2-NEU Positive
Drug: Taxotere — 75mg/m2 iv on day 1 of each 3 week cycle
  Arms: HER2-NEU Positive
Drug: Herceptin (HER2-neu positive patients only) — 4mg/kg iv (loading dose) followed by 2mg/kg iv weekly
  Arms: HER2-NEU Positive
Drug: capecitabine [Xeloda] — 825mg/m2 po bid on days 1-14 of each 3 week cycle
  Arms: HER2-NEU Negative
Drug: Taxotere — 75mg/m2 iv on day 1 of each 3 week cycle
  Arms: HER2-NEU Negative

SUMMARY:
This single arm study stratified patients into two treatment cohorts based on HER2-neu overexpression/amplification. Each cohort will be independently powered for the primary endpoint. The study will evaluate the efficacy, safety and impact on quality of life of treatment with oral Xeloda plus intravenous (iv) Taxotere (docetaxel). Patients with HER2-neu negative breast cancer will receive chemotherapy alone with oral Xeloda plus intravenous (iv) Taxotere (docetaxel). Patients with HER2-neu positive breast cancer, will receive the same chemotherapy in combination with intravenous (iv) Herceptin (trastuzumab). Patients will receive 3-weekly cycles of treatment with Xeloda (825mg/m2 oral administration [po] twice daily (bid) on days 1-14) + Taxotere (75mg/m2 iv on day 1). HER2-neu positive patients will also receive Herceptin (loading dose of 4mg/kg iv followed by 2mg/kg iv weekly). The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* women >=18 years of age;
* newly diagnosed;
* infiltrating (invasive) HER2-neu-negative or HER2-neu-positive breast cancer.

Exclusion Criteria:

* evidence of metastatic disease, except ipsilateral (same side) axillary lymph nodes;
* previous systemic or local primary treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2005-08; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- United States (33):
  - Los Angeles, California
  - Montebello, California
  - Palm Springs, California
  - San Diego, California
  - Farmington, Connecticut
  - Melbourne, Florida
  - Miami, Florida
  - Tamarac, Florida
  - Savannah, Georgia
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Alexandria, Louisiana
  - Scarborough, Maine
  - Baltimore, Maryland
  - Edina, Minnesota
  - Jefferson City, Missouri
  - Rolla, Missouri
  - St Louis, Missouri
  - Neptune City, New Jersey
  - Albuquerque, New Mexico
  - Santa Fe, New Mexico
  - New York, New York
  - Charlotte, North Carolina
  - Canton, Ohio
  - Pittsburgh, Pennsylvania
  - Pottsville, Pennsylvania
  - Charleston, South Carolina
  - Georgetown, South Carolina
  - Sumter, South Carolina
  - Memphis, Tennessee
  - Dallas, Texas
  - Burlington, Vermont
  - Abingdon, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- HER2-Neu Negative: Dose and route per treatment cycle (Q3W):
  Capecitabine: 825 mg/m2, orally, twice daily, days 1-14 Docetaxel: 75 mg/m2, IV infusion, day 1
  HER2-neu negative: capecitabine + docetaxel
  Duration: Four 3-week treatment cycles
- HER2-Neu Positive: Dose and route per treatment cycle (Q3W):
  Capecitabine: 825 mg/m2, orally, twice daily, days 1-14 Docetaxel: 75 mg/m2, IV infusion, day 1 Trastuzumab: loading dose 4 mg/kg, 90-min IV infusion; thereafter, 2 mg/kg, 30-min IV infusion, weekly
  HER2-neu positive: capecitabine + docetaxel + trastuzumab
  Duration: Four 3-week treatment cycles
Period: Overall Study
Arm/Group | HER2-Neu Negative | HER2-Neu Positive
Started | 123 | 34
Pathological Response | 101 | 28
Clinical Response | 122 | 34
Safety Population | 122 | 34
Quality of Life Population | 118 | 33
Postoperative | 98 | 27
Completed | 122 | 34
Not Completed | 1 | 0
Not completed — Randomized but not dosed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HER2-Neu Negative | HER2-Neu Positive | Total
Number analyzed (Participants) | 122 | 34 | 156
Age Continuous [Mean (Standard Deviation); unit: years] — Safety Population
  years | 51.0 (11.20) | 52.2 (9.36) | 51.3 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 34 | 156
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Assessed for Pathological Complete Response (pCR) Plus Near Complete (npCR) in Primary Breast Tumor at Time of Definitive Surgery
Description: Pathological complete response was defined as the absence of histological evidence of invasive breast cancer cells in the tissue specimen removed from the breast after 4 cycles of preoperative treatment. Near pCR (npCR) was defined as the presence of invasive tumor cells with a size of 5 mm or less in aggregate in the tissue specimen removed from the breast after 4 cycles of preoperative treatment. Only pathological assessments occurring prior to the first date of adjuvant treatment were included in the analysis of pCR rate.
Time Frame: at the time of definitive surgery; after four 3-week cycles (3-4 months)
Population: Pathological Response Evaluable Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2-Neu Negative | HER2-Neu Positive
Number analyzed (Participants) | 101 | 28
percentage of participants | 15.8 [9.7 to 25.4] | 50.0 [31.9 to 71.3]

2. Secondary Outcome: Percentage of Participants With Complete Pathological Response in the Primary Breast Tumor at the Time of Definitive Surgery
Description: Pathological complete response was defined as the absence of histological evidence of invasive breast cancer cells in the tissue specimen removed from the breast after 4 cycles of preoperative treatment.
Time Frame: at the time of definitive surgery; after four 3-week cycles (3-4 months)
Population: Pathological Response Evaluable Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2-Neu Negative | HER2-Neu Positive
Number analyzed (Participants) | 101 | 28
percentage of participants | 9.9 [5.1 to 18.1] | 35.7 [19.4 to 57.6]

3. Secondary Outcome: Percentage of Participants With Overall Clinical Response (Complete Response (CR) Plus Partial Response (PR))
Description: The best overall response in an individual patient, according to RECIST, during preoperative treatment was the best response recorded from the start of study treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the baseline assessment) or completion of preoperative treatment. Patients with CR or PR were considered responders. Patients with no tumor assessment after the start of study treatment were considered nonresponders.
Time Frame: post 2 and 4, 3-week cycles of treatment
Population: Evaluable Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2-Neu Negative | HER2-Neu Positive
Number analyzed (Participants) | 101 | 28
percentage of participants | 23.8 [18.6 to 35.9] | 23.5 [12.3 to 45.9]

4. Secondary Outcome: Percentage of Participants With Local Recurrence
Description: Local recurrence was defined as evidence of recurrent carcinoma in the same breast where it was diagnosed initially before preoperative treatment.
Time Frame: 30 - 1102 days
Population: Postoperative Response Evaluable Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2-Neu Negative | HER2-Neu Positive
Number analyzed (Participants) | 101 | 28
percentage of participants | 3.1 [0.6 to 8.7] | 3.7 [0.1 to 19.0]

5. Secondary Outcome: Participants With Disease-Free Survival
Description: Disease-free survival was defined as the time from date of surgery to date of first evidence of cancer recurrence in the breast (ie, local or distant recurrence or contra lateral disease) or death from any cause, whichever came first. Patients who were alive or withdrawn from the study and had no evidence of disease recurrence and for whom there was CRF evidence that evaluations had been made were censored at the date of the last clinical follow-up assessment when the patient was known to be disease free.
Time Frame: 30 - 1102 days
Population: The analysis was done on the Postoperative Response Evaluable Population.
Measure: Number; unit: participants
Arm/Group | HER2-Neu Negative | HER2-Neu Positive
Number analyzed (Participants) | 98 | 27
participants | 92 | 25

6. Secondary Outcome: Participants With Overall Survival
Description: Overall survival was defined as the time from date of start of study treatment to the date of death, regardless of the cause of death. Patients who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Patients without follow-up assessment were censored at the day of the last dose. Patients with no post-baseline information were censored at the start of study treatment.
Time Frame: 22 - 1191 days
Population: The analysis was done on the post-operative Response Evaluable Population.
Measure: Number; unit: participants
Arm/Group | HER2-Neu Negative | HER2-Neu Positive
Number analyzed (Participants) | 122 | 34
participants | 118 | 32

ADVERSE EVENTS:
Time Frame: Cycle 1, Cycle 2, Cycle 3, Cycle 4, at Surgery, and the month 1 visit during the postoperative follow-up period
Description: Intensity of AEs was graded according to the NCI CTCAE version 3.0 on a 5-point scale (grade 1 to 5), clinical laboratory parameters (hematology, chemistry, and urinalysis as clinically indicated), and vital signs.
Arm/Group | HER2-Neu Negative | HER2-Neu Positive
Serious Adverse Events (participants affected / at risk) | 15/122 | 7/34
Other Adverse Events (participants affected / at risk) | 121/122 | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HER2-Neu Negative (N=122) | HER2-Neu Positive (N=34)
febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1
Pneumonia (Infections and infestations) | 1 | 1
Catheter site cellulitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HER2-Neu Negative (N=122) | HER2-Neu Positive (N=34)
Nausea (Gastrointestinal disorders) | 57 | 19
Diarrhoea (Gastrointestinal disorders) | 51 | 19
Constipation (Gastrointestinal disorders) | 30 | 6
Stomatitis (Gastrointestinal disorders) | 18 | 14
Dyspepsia (Gastrointestinal disorders) | 22 | 6
Vomiting (Gastrointestinal disorders) | 24 | 4
Abdominal pain (Gastrointestinal disorders) | 11 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2
Haemorrhoids (Gastrointestinal disorders) | 4 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 57 | 21
Alopecia (Skin and subcutaneous tissue disorders) | 59 | 12
Rash (Skin and subcutaneous tissue disorders) | 29 | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 10 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 2
Erythema (Skin and subcutaneous tissue disorders) | 7 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 2
Fatigue (General disorders) | 62 | 20
Mucosal inflammation (General disorders) | 21 | 5
Oedema peripheral (General disorders) | 17 | 4
Pyrexia (General disorders) | 7 | 5
Pain (General disorders) | 6 | 6
Chest pain (General disorders) | 7 | 1
Chills (General disorders) | 5 | 4
Asthenia (General disorders) | 4 | 2
Chest discomfort (General disorders) | 2 | 2
Catheter site pain (General disorders) | 1 | 2
Headache (Nervous system disorders) | 20 | 4
Dysgeusia (Nervous system disorders) | 17 | 3
Neuropathy peripheral (Nervous system disorders) | 17 | 2
Paraesthesia (Nervous system disorders) | 8 | 3
Dizziness (Nervous system disorders) | 8 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 31 | 9
Anaemia (Blood and lymphatic system disorders) | 7 | 10
Insomnia (Psychiatric disorders) | 27 | 12
Anxiety (Psychiatric disorders) | 10 | 4
Depression (Psychiatric disorders) | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Vaginal infection (Infections and infestations) | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 10 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2
Lacrimation increased (Eye disorders) | 11 | 4
Eye irritation (Eye disorders) | 1 | 2
Flushing (Vascular disorders) | 6 | 2
Breast pain (Reproductive system and breast disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No